CLINICAL TRIAL: NCT06537817
Title: A Phase 1, First-in-Human, Randomized, Placebo-Controlled, Double-Blind Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses (SAD) and Multiple Ascending Doses (MAD) of Oral HT-4253 in Healthy Adults
Brief Title: Study to Evaluate HT-4253 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Halia Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: HT-4253-NHV-001
Record Dates: First submitted 2024-07-30; First posted 2024-08-05 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Normal Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HT-4253 (Experimental): Subjects will participate in 1 of 10 groups and receive single or multiple doses of HT-4253 or matching placebo. In each group 6 subjects will receive HT-4253.
  Interventions: Drug: HT-4253
- Placebo to match HT-4253 (Placebo Comparator): Subjects will participate in 1 of 10 groups and receive single or multiple doses of HT-4253 or matching placebo. In each group 2 subjects will receive matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HT-4253 — HT-4253 Single or Multiple doses administered orally as a tablet
  Arms: HT-4253
Drug: Placebo — Placebo to match HT-4253 Single or Multiple doses administered orally as a tablet
  Arms: Placebo to match HT-4253

SUMMARY:
The primary objectives of this study are to evaluate the safety and tolerability of HT-4253 when administered as single oral doses and multiple oral doses at escalating dose levels in healthy volunteer subjects.

The secondary objectives of this study are to characterize the pharmacokinetics (PK) and pharmacodynamics (PD) of HT-4253.

ELIGIBILITY:
Inclusion Criteria:

* Age is ≥ 18 years to 65 years
* Body mass index between 18 and 32 kg/m2
* Female subjects must be surgically sterile or post menopausal for at least 12 months. Females may be of child-bearing potential but must use double contraception.

Exclusion Criteria:

* Any clinically significant central nervous system, cardiac, pulmonary, renal, gastrointestinal, endocrinological, respiratory, or metabolic conditions (or history), or other pathological or physiological conditions,
* History of suicidal behavior and/or ongoing suicidal ideation per C-SSRS evaluation when screening
* Use of any medications, including prescription, over-the-counter (OTC) medications, vitamins, herbal preparations, and supplements
* Positive drug screen or alcohol breath tests
* History of heavy smoking more than 10 cigarettes a day or the tobacco/nicotine equivalent within 3 months of Screening or refuses to abstain from tobacco or nicotine-containing products throughout the duration of the study
* Clinical significant abnormalities in laboratory test results
* Chronic or current active infectious disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single and multiple ascending doses of oral HT-4253 in healthy adults | up to 6 weeks
  Incidence of adverse events (AEs)
To evaluate the safety and tolerability of single and multiple ascending doses of oral HT-4253 in healthy adults | up to 6 weeks
  Serious adverse events (SAEs)
To evaluate the safety and tolerability of single and multiple ascending doses of oral HT-4253 in healthy adults | up to 6 weeks
  Treatment-related adverse events (TRAEs)
To evaluate the safety and tolerability of single and multiple ascending | up to 6 weeks
  Incidence of withdrawals due to AE

SECONDARY OUTCOMES:
To evaluate the plasma pharmacokinetics (PK) of single and multiple ascending doses of oral HT-4253 in healthy adults | up to 6 weeks
  Maximum plasma concentration (Cmax)
To evaluate the plasma pharmacokinetics (PK) of single and multiple ascending doses of oral HT-4253 in healthy adults | up to 6 weeks
  Area under the concentration-time curve (AUC)
To evaluate the plasma pharmacokinetics (PK) of single and multiple ascending doses of oral HT-4253 in healthy adults | up to 6 weeks
  Elimination half-life (t1/2) plasma concentration of HT-4253
To evaluate the plasma pharmacokinetics (PK) of single and multiple ascending doses of oral HT-4253 in healthy adults | up to 6 weeks
  Trough plasma concentration of HT-4253

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No